CLINICAL TRIAL: NCT01287143
Title: Beyond Intuition: Quantifying and Understanding the Signs and Symptoms of Fever
Brief Title: Quantifying and Understanding the Signs and Symptoms of Fever
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 110083; 11-CC-0083
Record Dates: First submitted 2011-01-29; First posted 2011-02-01 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-08-09

CONDITIONS: Fever
Keywords: Fever; Signs and Symptoms; Febrile Assessment Tool (FAST)
MeSH Terms: conditions — Fever; Signs and Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Background:

- Fever is a common symptom of illness, but it can involve many signs (a signal that something is not right in the body that can be seen by others, such as vomiting) and symptoms (a signal that something is not right in the body that are felt only by the person, such as pain) that may differ depending on the type of illness involved. Researchers are interested in studying individuals who have a fever to examine how often these signs and symptoms are experienced by patients.

Objectives:

- To identify and evaluate the signs and symptoms of fever and examine their frequency in individuals who have fever.

Eligibility:

- Individuals at least 8 years of age who are admitted to the NIH Clinical Center and have a fever (body temperature of at least 38 degrees Celsius/100.4 degrees Fahrenheit).

Design:

* Participants will be screened upon admission to the NIH Clinical Center.
* Researchers will review the Clinical Center admission records.
* Participants will complete a 15- to 20-minute survey with questions about how they are feeling and what symptoms they have experienced before, during and after an episode of fever.

DETAILED DESCRIPTION:
Background:

Fever is one of the most prevalent signs in hospitalized patients, signaling the activation of the immune system.

There is little empiric evidence related to symptoms or signs that accompany changes in body temperature.

Understanding the nature, timing and relationship of patient signs and symptoms of fever will provide insight into the febrile process and guide more informed treatment.

Objectives:

The protocol is divided into two phases:

Phase I

-To develop and implement a simple clinical tool for assessing and documenting patient-reported signs and symptoms of fever.

Phase II

-To describe the prevalence and relationship of signs and symptoms that accompanies a febrile state and related patterns of change over time.

Eligibility:

Phase I

* Adult and pediatric medical-surgical patients hospitalized at the Clinical Center admitted to 3NE (oncology/ transplant), 3NW (surgical oncology) and 1NW (pediatric).
* Age greater than or equal to 8 years old
* Understand and speak English

Phase II

* Inpatients admitted to the Clinical Research Center
* Age greater than or equal to 8 years old.

Design:

Phase I

-Descriptive study involving qualitative interviews and chart reviews from medical surgical inpatients. Two types of interviews with two different sets of patients will be conducted. The maximum number of research participants for this phase will be 65. The final sample size will be determined based on the point of saturation, defined as four consecutive interviews during which no new signs or symptoms associated with fever are identified. The second set of interviews will involve 20 to 30 new research participants, including at least 5 patients less than 18 years of age who will review a list of signs and symptoms of fever for comprehension and clarity to inform the final list and determine the terminology to be used in the FAST.

Study of the Febrile Assessment Tool (FAST)

-Test of the FAST in 120 patients. Before placing the FAST in the electronic record (Clinical Research Information System-CRIS) this new assessment tool will be used in approximately 120 patients during routine vital sign measurements. Patients admitted to the surgical oncology unit (3NW) will be consented and followed with collection of the FAST assessments

Education Implementation

* Inform nursing staff of the background, content and procedures for using the Febrile Assessment Tool (FAST)
* Educational interim will last 4 weeks

Phase II

* Approximately 2 months or at the discretion of the PI after FAST education
* Descriptive study involving chart review from unidentified inpatients. The sample size will be a maximum of 500.

ELIGIBILITY:
* INCLUSION CRITERIA PHASE I:

Adult and pediatric medical-surgical patients hospitalized in the Clinical Center, NIH admitted to 3NE (oncology/ transplant), 3NW (surgical oncology) and 1NW (pediatrics).

Oriented to person, time and place at time of interview

Active fever (body temperature greater than or equal to 38.0 Celsius), treated or untreated, within the last 12 hours.

Willingness to participate in a short interview (15-20 minutes) about their symptoms

Understands and speaks English

Age 8 years and older

INCLUSION CRITERIA FOR STUDY OF FEBRILE ASSESSMENT TOOL:

Adult (18 years of age or greater) medical-surgical patients hospitalized at the Clinical Center and admitted to 3NW.

Oriented to person, time and place at time of admission

Willingness to be asked about their symptoms of fever during vital signs assessment

Understands and speaks English

INCLUSION CRITERIA PHASE II:

Inpatients admitted to the Clinical Center

Age 8 years and older

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-01-13; Study Completion 2017-08-09

PRIMARY OUTCOMES:
Symptoms of fever | Throughout in patient admission

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ames, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Laupland KB. Fever in the critically ill medical patient. Crit Care Med. 2009 Jul;37(7 Suppl):S273-8. doi: 10.1097/CCM.0b013e3181aa6117. PMID 19535958
- [Background] Chesnutt BK, Zamora MR, Kleinpell RM. Blood cultures for febrile patients in the acute care setting: too quick on the draw? J Am Acad Nurse Pract. 2008 Nov;20(11):539-46. doi: 10.1111/j.1745-7599.2008.00356.x. PMID 19128337
- [Background] Bor DH, Makadon HJ, Friedland G, Dasse P, Komaroff AL, Aronson MD. Fever in hospitalized medical patients: characteristics and significance. J Gen Intern Med. 1988 Mar-Apr;3(2):119-25. doi: 10.1007/BF02596115. PMID 3357068
- [Derived] Ames NJ, Powers JH, Ranucci A, Gartrell K, Yang L, VanRaden M, Leidy NK, Wallen GR. A systematic approach for studying the signs and symptoms of fever in adult patients: the fever assessment tool (FAST). Health Qual Life Outcomes. 2017 Apr 27;15(1):84. doi: 10.1186/s12955-017-0644-6. PMID 28449675